CLINICAL TRIAL: NCT05413486
Title: Circadian Disturbances in People With Mental Disease
Brief Title: Sleep, Obesity and Mental Disease - Biological Markers for the Evaluation of Circadian Rhythmicity
Acronym: SOMBER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: Steno Diabetes Center Odense (Other); Region of Southern Denmark (Other); Rigshospitalet, Denmark (Other); University of Southern Denmark (Other); Odense University Hospital (Other); Odense Patient Data Explorative Network (Other)
Responsible Party: Sponsor
Other Study IDs: 21/61643
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Bipolar Disorder; Schizophrenia; Obesity; Circadian Rhythm Disorders
Keywords: Obesity; Schizophrenia; Bipolar Disorder; Circadian disturbances; Hair follicles; Clock genes; Cortisol; Melatonin; Sleep; mRNA
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia; Obesity; Chronobiology Disorders | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples tested for cortisol and melatonin content
  Hair follicle samples, tested for expression of specifically targeted clock genes.*
  *Hair follicles will be analyzed for gene expression using the PCR-based method real-time quantitative polymerase chain reaction (RT-qPCR). Investigators only obtain expression levels of genes targeted with specific commercially available primers. Therefore, NO information about the mRNA sequence or potential sequence variations in the selected set of genes will be investigated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- SCH, OB: People with obesity (BMI > 30 kg/m2) and a medical diagnosis of schizophrenia spectrum disorder.
  Interventions: Other: Observational
- BD, OB: People with obesity (BMI > 30 kg/m2) and a medical diagnosis of bipolar spectrum disorder.
  Interventions: Other: Observational
- Control, OB: Control group with obesity. People with obesity (BMI > 30 kg/m2) without psychiatric disease or sleep disorders.
  Interventions: Other: Observational
- Control, non-OB: Normal weight (BMI 18.5 - 25kg/m2) control group without psychiatric disease.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Exposure is defined by group affiliation i.e., Bipolar disorder vs. schizophrenia vs. no disease. Likewise with obesity vs. normal weight.
  Biological markers of daytime-circadian rhythmicity is compared across disease and weight groups.

SUMMARY:
Introduction

16.8% of the Danish adult population are obese (Body Mass Index> 30 kg / m2). Obesity increases the risk of lifestyle diseases such as type-2 diabetes and non-alcoholic fatty liver. People with mental illness have an increased risk of developing obesity. Both obesity and certain mental disorders (bipolar disorder and schizophrenia) are associated with circadian rhythm disorders. Clinically, this may manifest as reduced sleep quality, depressive symptoms and increased fatigue, but also deregulation of a wide range of bodily processes subject to the circadian rhythm.

In circadian rhythm disorders, the pattern of how mRNA of specific 'clock genes' is expressed in the cell may be affected. These clock genes are associated with obesity, bipolar disorder and schizophrenia. Despite the clear indications of an interplay between mental illness, obesity and circadian rhythm disorders, the relationship between these illnesses are largely unexplored.

Aim

The aim of this study is to investigate circadian disturbances in people with and without obesity, as well as people with obesity and a comorbid diagnosis of either schizophrenia or bipolar disorder.

Methods

The study population will consist of:

1. People with obesity and schizophrenia (N=22)
2. People with obesity and bipolar disorder (N=22)
3. People with obesity without psychiatric disease (N=22)
4. People with BMI 18.5 - 25kg/m2 and no psychiatric disease (N=20)

Study Procedure

Participants will visit the clinic 2 times. At each visit participants fill in questionnaires and perform physical tests. Between visit 1 and 2, participants will over a 2-day period (at-home), collect biological samples (Four hair- and six saliva samples per day). In addition, participants will wear accelerometers and continuous glucose monitors (CGMs) for a total of 8 days, including the 2-day sampling period.

Sampled hair follicles are analyzed for relative expression of clock gene mRNA. Saliva is analyzed for cortisol- and melatonin content. The four participants groups are analyzed and compared on daytime variation in mRNA expression, cortisol- and melatonin concentration, and body temperature.

Perspectives

A comparison of patient groups presenting with mental disease, obesity and circadian disturbances may provide new insight into the association between these diseases.

DETAILED DESCRIPTION:
Background

Obesity (30 ≥ kg/m2) is a major global health challenge. Worldwide obesity has nearly tripled since 1975 (WHO, 2021) and is projected to continue to rise throughout western society (OECD, 2017).

Obesity increases the risk of type-2 diabetes (T2D), obstructive sleep apnea (OSA), non-alcoholic fatty liver disease (NAFLD), hypertension, osteoarthritis, polycystic ovary syndrome and several other conditions (George et al., 2018; Luque-Ramirez et al., 2014; Mainous, Tanner, Jo, & Anton, 2016). Mortality is significantly increased, and a person with class III obesity (BMI > 40kg/m2) is predicted to live ten years shorter than a normal-weight person of same age (Finkelstein, Brown, Wrage, Allaire, & Hoerger, 2010). People with obesity have more days of sick leave, experience social disadvantages (Hernaes, Andersen, Norheim, & Vage, 2015) and report an overall poorer health-related quality of life compared to non-obese people (Kolotkin & Andersen, 2017).

Obesity and mental disease:

Mental disease is associated with increased risk of obesity. Obesity is approximately two and three times as prevalent in people with bipolar disorders and schizophrenia spectrum disorder compared to people without mental disease, respectively (Annamalai, Kosir, & Tek, 2017; Chao, Wadden, & Berkowitz, 2019; Sicras, Rejas, Navarro, Serrat, & Blanca, 2008). Many commonly used antipsychotic drugs induces weight gain with a magnitude ranging from neutral in some drugs to +5.3 kg in olanzapine (Vancampfort et al., 2015). Antipsychotic-induced weight changes depend of the underlying disease (Moteshafi, Zhornitsky, Brunelle, & Stip, 2012). Many mental diseases are associated with higher calorie intake, poorer food quality (Manu et al., 2015) and lower levels of physical activity (Schuch et al., 2017; Vancampfort et al., 2017).

Obesity, mental disease and circadian disturbances:

The human body adapts cellular, physiological, and behavioral rhythms to the 24-hour light cycle. Disturbing the normal circadian rhythms have dramatic consequences on many health issues ranging from cardiovascular disease to cancer (Morris, Purvis, Hu, & Scheer, 2016; Stevens, Brainard, Blask, Lockley, & Motta, 2014). A sleep pattern concordant with the diurnal rhythm is crucial for maintaining normal body weight. Sleeping incoherently with the circadian-defined sleep hours thus independently associates with overweight and obesity, increasing the relative risk by 31% and 96% respectively (McFadden, Jones, Schoemaker, Ashworth, & Swerdlow, 2014). In people with schizophrenia and bipolar disorders almost all measures of sleep quality and physiological sleep patterns are disturbed, even when their disease is considered well-treated (Meyer et al., 2020).

In human cells, circadian clocks are composed of a set of proteins that generate self-sustained circadian oscillation through positive and negative transcriptional/translational feedback loops. The human circadian clock entails a range of 'clock genes'. For example: The 'Period' genes (per1 and per2) are both parts of the circadian feedback loop. Mice models knocked out for per1/2 completely lacks a diurnal rhythm and gain more weight following a high-fat diet (Dallmann & Weaver, 2010). Dysregulation of per1, per2 and other clock genes have been linked to psychiatric disorders, including depression, schizophrenia and bipolar disorders (Charrier, Olliac, Roubertoux, & Tordjman, 2017).

Altogether disturbance in clock-gene and hormonal rhythmicity might be an important link between mental disease, sleep disturbance and obesity. Sleep disturbances are potentially treatable. Accordingly, restoration of sleep patterns might be a possible target to prevent weight gain and obesity in this group of patients.

Study aim:

To evaluate biological markers of disturbed circadian rhythm in people with obesity and schizophrenia or bipolar disorder.

Overall hypotheses:

People with obesity and schizophrenia or bipolar disorder has disturbed circadian rhythms compared to controls without mental disease.

Methods

Study design:

This will be a single-center case-control study with repeated measures.

Study Population:

The study population will consist of four groups:

1. People with BMI > 30 kg/m2 and schizophrenia spectrum disorder (N=22)
2. People with BMI > 30 kg/m2 and bipolar spectrum disorder (N=22)
3. People with BMI > 30 kg/m2 without psychiatric disease or sleep disorders (N=22)
4. People with BMI 18.5 - 25kg/m2 and no psychiatric disease or sleep disorders (N=20)

Exclusion criterion:

• Participants taking oral supplements of melatonin are excluded if pausing is deemed inappropriate.

Study Procedure:

Participants will visit the clinic two times. Between visits, participants will collect biological samples and data relevant to understanding circadian rhythms over a 2-day period. In addition participants will wear accelerometers and continuous glucose monitors (CGMs) for a total of 8 days.

Clinical visit 1:

During the first clinical visit, a short (<10 min) test battery will be administered. This includes tests of gait function, handgrip strength and balance. In addition weight, height, waist- and hip circumference and body composition (by bioimpedance) are measured. After tests, a short questionnaire is administered.

Finally, body worn sensors (accelerometers and CGMs) are mounted, and the participant is given thorough instruction on how to record dietary intake and perform biological sampling (hair and saliva samples). The two sampling days will, when possible, be placed immediately following clinical visit 1 and at least within 5 days.

At-home testing:

During test day 1 and 2, participants will collect saliva samples ~6 times (depended on bed time) per day and hair samples 4 times per day and record their body temperature and dietary food intake (see "data collection" below). Participants will each day receive home visits from the project manager. If possible, visits will be scheduled around noon in order to aid participants with mid-day sampling. Visits are scheduled to take <20 minutes. During visits, the project manager will administer a short questionnaire on media device usage and sleep environment light exposure.

Clinical visit 2:

Following the two sampling days, participants will again meet at the clinic. During this visit, remaining test equipment and samples are handed over. Afterwards, the patient fills in the Morningness-Eveningness Questionnaire (MEQ). In addition, the test leader will perform a short interview (~10 min) in which participants are asked to rate their experience. If the participant have not been screened for sleep apnea recently (<6months), a time for respiratory sleep monitoring will be scheduled.

Data handling and analyses:

Data will be hosted and handled in accordance with Danish law and regulation. All data Files will be kept for 5 years following study conclusion and subsequently anonymized or deleted.

Statistics:

Disturbances in circadian rhythm will be analyzed by multi-level longitudinal analyses comparing findings between study groups (BMI >30 kg/m2, ≤25 kg/m2, with and without mental disease) adjusted for gender and age. Associations between circadian regulated variables (hormones, temperature, glucose levels and gene expression) will be investigated by correlational analysis.

Power calculation:

Being explorative in nature, there is insufficient data to conduct a candid power-calculation. However recent studies detected significant differences in clock-gene expression between people with and without sleep disturbances with 14 to 20 people in each study group (Canales et al., 2019; Zhanfeng, Hechun, Zhijun, Hongyu, & Zhou, 2019).

Information from patient registries:

After consent is signed, patient journals will be reviewed for information on age, gender, socioeconomic status, medication status and the presence of psychiatric diagnoses (Bi-polar, schizophrenia and depression), medication history and obesity-related disease prevalence.

Financing and insurance:

This is an investigator initiated research project. The Project received 913.000 kr.- from Region Syddanmarks pulje for Fri og Strategisk Forskning 2021 to cover running expenses. Study funds are placed on a dedicated account and the account number has been disseminated to the Regional Committee on Health Research Ethics for Southern Denmark. The investigators or The Department of Medicine, University Hospital South West Jutland have no financial gain regarding the study and have no conflict of interest that could be perceived as prejudicing the impartiality of this study. The patients will not receive payment but reimbursement of travel expenses can be made.

Side effects, risks and complications:

The study is designed to minimize inconvenience by employing a relative short list of outcomes requiring active participant involvement. Moreover, participant work loads are minimized through the use of digital solutions. Participants are not required to record sleep or food diaries and do not need to weigh food items as these are recorded by digital camera.

There are no known risks associated with present study procedure. Participants are informed of potential discomfort when plucking hairs or when mounting the CGM and that some may experience poorer sleep quality when sleeping with the CRM instrument. Participants are encouraged to report any adverse events experienced during or following the study procedure. In case of injury participant are instructed to report their case to the Danish national patient compensation scheme (http://www.patientforsikringen.dk), also linked in the participant information.

Perspectives

Comparative data on patient groups presenting with mental disease, obesity and circadian disturbances may help elucidate the association between these diseases. If circadian disturbances are more pronounced in people with obesity and schizophrenia or bipolar disorder, compared to people with obesity and no mental disease, this highlights the need for treatment effective in normalizing sleep patterns in these patient groups.

ELIGIBILITY:
Inclusion Criteria:

Fulfilling the criteria for one of the four study groups:

* People with BMI > 30 kg/m2 and schizophrenia spectrum disorder (N=22)
* People with BMI > 30 kg/m2 and bipolar disorder spectrum disorder (N=22)
* People with BMI > 30 kg/m2 without psychiatric disease or sleep disorders (N=22)
* People with BMI 18.5 - 25kg/m2 and no psychiatric disease or sleep disorders (N=20)

Exclusion Criteria:

* Participants taking oral supplements of melatonin are excluded if pausing is deemed inappropriate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants may be recruited by two pathways:
  1. Referral through psychiatric treatment units*
  2. Referral through the South Danish Obesity initiative (SDOI)
     * In addition to local treatment clinics this includes the following collabarative networks: OPT (Opsøgende Psykoseteam (english: outreach Psychosis team)), OPUS (Opsøgende Psykoseteam for Unge med Skizofreni (english: outreach Psychosis team for young adults with schizophrenia) and Psykinfo (a mental health information service in the Region of Southern Denmark).
  A third pathway is available for healthy controls: Posters are placed in libraries, groceries and educational facilities and by advertising in select local Facebook groups, especially targeting young (>30 years) adults.
  While no formal exclussion criteria is presented regarding symptom severity. Health workers at psychiatric treatment units and SDOI will only refer participants with a high propability of completing the examination program.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Daytime Circadian variation in clock gene mRNA expression | for two full consecutive days participant will pluck hairs and place the hair root in a dissolution buffer. Participants will each collect 4 samples per day: immediately after waking, and every 6th preceding hour, including immediately before bed.
  Relative amount of different clock gene mRNA, compared to housekeeping gene

SECONDARY OUTCOMES:
Daytime Circadian variation in saliva melatonin concentration | for two full consecutive days participant will collect saliva samples. Participants will each collect ~6 samples per day: immediately after waking, 6 and 12 hours after waking and every 2 hours until bedtime, including a sample immediately before bed.
  Saliva samples are analyzed for melatonin concentration throughout the day.
Daytime Circadian variation in saliva cortisol concentration | for two full consecutive days participant will collect saliva samples. Participants will each collect ~6 samples per day: immediately after waking, 6 and 12 hours after waking and every 2 hours until bedtime, including a sample immediately before bed.
  Saliva samples are analyzed for cortisol concentration throughout the day.

OTHER OUTCOMES:
Sleep amount and quality | Participant will wear accelerometers for 8 consecutive days. The two self-sampling days and an additional 6 days.
  assessed by accelerometry (placement: right thigh and non-dominant wrist)
Continous glucose monitoring | Participant will wear glucose monitors for 8 consecutive days. The two self-sampling days and an additional 6 days.
  glucose levels are monitored using a body-worn monitor (freestyle libre)
Dietary intake and timing | Participants will record dietary items for two consecutive days (the two self-sampling days)
  Timing of food consumption, total caloric intake and caloric distribution (fat, protein, carbohydrates) will be estimated using a digital food diary

CONTACTS AND LOCATIONS:
Overall Officials: Claus B Juhl, Principal Investigator — University Hospital South West Jutland, Department of Endocrinology
Locations (1):
- Hospital South West Jutland, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: No
Sharing of IPD is under current Danish law not feasible.

REFERENCES:
- [Background] Mainous AG 3rd, Tanner RJ, Jo A, Anton SD. Prevalence of Prediabetes and Abdominal Obesity Among Healthy-Weight Adults: 18-Year Trend. Ann Fam Med. 2016 Jul;14(4):304-10. doi: 10.1370/afm.1946. PMID 27401417
- [Background] George ES, Roberts SK, Nicoll AJ, Reddy A, Paris T, Itsiopoulos C, Tierney AC. Non-alcoholic fatty liver disease patients attending two metropolitan hospitals in Melbourne, Australia: high risk status and low prevalence. Intern Med J. 2018 Nov;48(11):1369-1376. doi: 10.1111/imj.13973. PMID 29845719
- [Background] Luque-Ramirez M, Marti D, Fernandez-Duran E, Alpanes M, Alvarez-Blasco F, Escobar-Morreale HF. Office blood pressure, ambulatory blood pressure monitoring, and echocardiographic abnormalities in women with polycystic ovary syndrome: role of obesity and androgen excess. Hypertension. 2014 Mar;63(3):624-9. doi: 10.1161/HYPERTENSIONAHA.113.02468. Epub 2013 Dec 9. PMID 24324038
- [Background] Finkelstein EA, Brown DS, Wrage LA, Allaire BT, Hoerger TJ. Individual and aggregate years-of-life-lost associated with overweight and obesity. Obesity (Silver Spring). 2010 Feb;18(2):333-9. doi: 10.1038/oby.2009.253. Epub 2009 Aug 13. PMID 19680230
- [Background] Hernaes UJ, Andersen JR, Norheim OF, Vage V. Work participation among the morbidly obese seeking bariatric surgery: an exploratory study from Norway. Obes Surg. 2015 Feb;25(2):271-8. doi: 10.1007/s11695-014-1333-8. PMID 24980085
- [Background] Kolotkin RL, Andersen JR. A systematic review of reviews: exploring the relationship between obesity, weight loss and health-related quality of life. Clin Obes. 2017 Oct;7(5):273-289. doi: 10.1111/cob.12203. Epub 2017 Jul 10. PMID 28695722
- [Background] Heltberg A, Andersen JS, Sandholdt H, Siersma V, Kragstrup J, Ellervik C. Predictors of undiagnosed prevalent type 2 diabetes - The Danish General Suburban Population Study. Prim Care Diabetes. 2018 Feb;12(1):13-22. doi: 10.1016/j.pcd.2017.08.005. Epub 2017 Sep 28. PMID 28964672
- [Background] Peromaa-Haavisto P, Tuomilehto H, Kossi J, Virtanen J, Luostarinen M, Pihlajamaki J, Kakela P, Victorzon M. Prevalence of Obstructive Sleep Apnoea Among Patients Admitted for Bariatric Surgery. A Prospective Multicentre Trial. Obes Surg. 2016 Jul;26(7):1384-90. doi: 10.1007/s11695-015-1953-7. PMID 26559426
- [Background] Spurr S, Bally J, Hill P, Gray K, Newman P, Hutton A. Exploring the Prevalence of Undiagnosed Prediabetes, Type 2 Diabetes Mellitus, and Risk Factors in Adolescents: A Systematic Review. J Pediatr Nurs. 2020 Jan-Feb;50:94-104. doi: 10.1016/j.pedn.2019.09.025. Epub 2019 Nov 28. PMID 31786470
- [Background] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183
- [Background] Laiteerapong N, Ham SA, Gao Y, Moffet HH, Liu JY, Huang ES, Karter AJ. The Legacy Effect in Type 2 Diabetes: Impact of Early Glycemic Control on Future Complications (The Diabetes & Aging Study). Diabetes Care. 2019 Mar;42(3):416-426. doi: 10.2337/dc17-1144. Epub 2018 Aug 13. PMID 30104301
- [Background] Stefan N, Haring HU, Hu FB, Schulze MB. Metabolically healthy obesity: epidemiology, mechanisms, and clinical implications. Lancet Diabetes Endocrinol. 2013 Oct;1(2):152-62. doi: 10.1016/S2213-8587(13)70062-7. Epub 2013 Aug 30. PMID 24622321
- [Background] Chao AM, Wadden TA, Berkowitz RI. Obesity in Adolescents with Psychiatric Disorders. Curr Psychiatry Rep. 2019 Jan 19;21(1):3. doi: 10.1007/s11920-019-0990-7. PMID 30661128
- [Background] Annamalai A, Kosir U, Tek C. Prevalence of obesity and diabetes in patients with schizophrenia. World J Diabetes. 2017 Aug 15;8(8):390-396. doi: 10.4239/wjd.v8.i8.390. PMID 28861176
- [Background] Sicras A, Rejas J, Navarro R, Serrat J, Blanca M. Metabolic syndrome in bipolar disorder: a cross-sectional assessment of a Health Management Organization database. Bipolar Disord. 2008 Jul;10(5):607-16. doi: 10.1111/j.1399-5618.2008.00599.x. PMID 18657245
- [Background] Vancampfort D, Stubbs B, Mitchell AJ, De Hert M, Wampers M, Ward PB, Rosenbaum S, Correll CU. Risk of metabolic syndrome and its components in people with schizophrenia and related psychotic disorders, bipolar disorder and major depressive disorder: a systematic review and meta-analysis. World Psychiatry. 2015 Oct;14(3):339-47. doi: 10.1002/wps.20252. PMID 26407790
- [Background] Baldessarini RJ. Comparing tolerability of olanzapine in schizophrenia and affective disorders: a meta-analysis. Drug Saf. 2012 Dec 1;35(12):1183; author reply 1183-4. doi: 10.2165/11641670-000000000-00000. No abstract available. PMID 23137152
- [Background] Manu P, Dima L, Shulman M, Vancampfort D, De Hert M, Correll CU. Weight gain and obesity in schizophrenia: epidemiology, pathobiology, and management. Acta Psychiatr Scand. 2015 Aug;132(2):97-108. doi: 10.1111/acps.12445. Epub 2015 May 27. PMID 26016380
- [Background] Schuch F, Vancampfort D, Firth J, Rosenbaum S, Ward P, Reichert T, Bagatini NC, Bgeginski R, Stubbs B. Physical activity and sedentary behavior in people with major depressive disorder: A systematic review and meta-analysis. J Affect Disord. 2017 Mar 1;210:139-150. doi: 10.1016/j.jad.2016.10.050. Epub 2016 Nov 29. PMID 28033521
- [Background] Vancampfort D, Firth J, Schuch FB, Rosenbaum S, Mugisha J, Hallgren M, Probst M, Ward PB, Gaughran F, De Hert M, Carvalho AF, Stubbs B. Sedentary behavior and physical activity levels in people with schizophrenia, bipolar disorder and major depressive disorder: a global systematic review and meta-analysis. World Psychiatry. 2017 Oct;16(3):308-315. doi: 10.1002/wps.20458. PMID 28941119
- [Background] Lucassen EA, Coomans CP, van Putten M, de Kreij SR, van Genugten JH, Sutorius RP, de Rooij KE, van der Velde M, Verhoeve SL, Smit JW, Lowik CW, Smits HH, Guigas B, Aartsma-Rus AM, Meijer JH. Environmental 24-hr Cycles Are Essential for Health. Curr Biol. 2016 Jul 25;26(14):1843-53. doi: 10.1016/j.cub.2016.05.038. Epub 2016 Jul 14. PMID 27426518
- [Background] Morris CJ, Purvis TE, Hu K, Scheer FA. Circadian misalignment increases cardiovascular disease risk factors in humans. Proc Natl Acad Sci U S A. 2016 Mar 8;113(10):E1402-11. doi: 10.1073/pnas.1516953113. Epub 2016 Feb 8. PMID 26858430
- [Background] Stevens RG, Brainard GC, Blask DE, Lockley SW, Motta ME. Breast cancer and circadian disruption from electric lighting in the modern world. CA Cancer J Clin. 2014 May-Jun;64(3):207-18. doi: 10.3322/caac.21218. Epub 2013 Dec 24. PMID 24604162
- [Background] McFadden E, Jones ME, Schoemaker MJ, Ashworth A, Swerdlow AJ. The relationship between obesity and exposure to light at night: cross-sectional analyses of over 100,000 women in the Breakthrough Generations Study. Am J Epidemiol. 2014 Aug 1;180(3):245-50. doi: 10.1093/aje/kwu117. Epub 2014 May 29. PMID 24875371
- [Background] Meyer N, Faulkner SM, McCutcheon RA, Pillinger T, Dijk DJ, MacCabe JH. Sleep and Circadian Rhythm Disturbance in Remitted Schizophrenia and Bipolar Disorder: A Systematic Review and Meta-analysis. Schizophr Bull. 2020 Sep 21;46(5):1126-1143. doi: 10.1093/schbul/sbaa024. PMID 32154882
- [Background] Dallmann R, Weaver DR. Altered body mass regulation in male mPeriod mutant mice on high-fat diet. Chronobiol Int. 2010 Jul;27(6):1317-28. doi: 10.3109/07420528.2010.489166. PMID 20653457
- [Background] Charrier A, Olliac B, Roubertoux P, Tordjman S. Clock Genes and Altered Sleep-Wake Rhythms: Their Role in the Development of Psychiatric Disorders. Int J Mol Sci. 2017 Apr 29;18(5):938. doi: 10.3390/ijms18050938. PMID 28468274
- [Background] Peschke E, Bahr I, Muhlbauer E. Melatonin and pancreatic islets: interrelationships between melatonin, insulin and glucagon. Int J Mol Sci. 2013 Mar 27;14(4):6981-7015. doi: 10.3390/ijms14046981. PMID 23535335
- [Background] Lewis P, Oster H, Korf HW, Foster RG, Erren TC. Food as a circadian time cue - evidence from human studies. Nat Rev Endocrinol. 2020 Apr;16(4):213-223. doi: 10.1038/s41574-020-0318-z. Epub 2020 Feb 13. PMID 32055029
- [Background] Bogdan A, Bouchareb B, Touitou Y. Ramadan fasting alters endocrine and neuroendocrine circadian patterns. Meal-time as a synchronizer in humans? Life Sci. 2001 Feb 23;68(14):1607-15. doi: 10.1016/s0024-3205(01)00966-3. PMID 11263673
- [Background] Harada T, Hirotani M, Maeda M, Nomura H, Takeuchi H. Correlation between breakfast tryptophan content and morning-evening in Japanese infants and students aged 0-15 yrs. J Physiol Anthropol. 2007 Mar;26(2):201-7. doi: 10.2114/jpa2.26.201. PMID 17435366
- [Background] van Faassen M, Bischoff R, Kema IP. Relationship between plasma and salivary melatonin and cortisol investigated by LC-MS/MS. Clin Chem Lab Med. 2017 Aug 28;55(9):1340-1348. doi: 10.1515/cclm-2016-0817. PMID 27997348
- [Background] Rasmussen MGB, Pedersen J, Olesen LG, Brage S, Klakk H, Kristensen PL, Brond JC, Grontved A. Short-term efficacy of reducing screen media use on physical activity, sleep, and physiological stress in families with children aged 4-14: study protocol for the SCREENS randomized controlled trial. BMC Public Health. 2020 Mar 23;20(1):380. doi: 10.1186/s12889-020-8458-6. PMID 32293374
- [Background] Ancoli-Israel S, Cole R, Alessi C, Chambers M, Moorcroft W, Pollak CP. The role of actigraphy in the study of sleep and circadian rhythms. Sleep. 2003 May 1;26(3):342-92. doi: 10.1093/sleep/26.3.342. PMID 12749557
- [Background] Zhanfeng N, Hechun X, Zhijun Z, Hongyu X, Zhou F. Regulation of Circadian Clock Genes on Sleep Disorders in Traumatic Brain Injury Patients. World Neurosurg. 2019 Oct;130:e475-e486. doi: 10.1016/j.wneu.2019.06.122. Epub 2019 Jun 25. PMID 31252075
- [Background] Canales MT, Holzworth M, Bozorgmehri S, Ishani A, Weiner ID, Berry RB, Beyth RJ, Gumz M. Clock gene expression is altered in veterans with sleep apnea. Physiol Genomics. 2019 Mar 1;51(3):77-82. doi: 10.1152/physiolgenomics.00091.2018. Epub 2019 Jan 18. PMID 30657733
- [Background] Danish Board on Health, Danskernes sundhed - Den Nationale Sundhedsprofil 2021 [Danish Health - The National Health Profile 2021]. 2022. available from: https://www.sst.dk/da/Udgivelser/2022/Danskernes-sundhed
- [Background] OECD [Organization for Economic Co-operation and Development]. Obesity update 2017. Available from: https://www.oecd.org/health/obesity-update.htm
- [Derived] Kolind ME, Kruse R, Petersen AS, Larsen CS, Bak LK, Hojlund K, Beier CP, Stenager E, Juhl CB. Investigating the role of obesity, circadian disturbances and lifestyle factors in people with schizophrenia and bipolar disorder: Study protocol for the SOMBER trial. PLoS One. 2024 Jul 8;19(7):e0306408. doi: 10.1371/journal.pone.0306408. eCollection 2024. PMID 38976708